CLINICAL TRIAL: NCT06038565
Title: Comparing Regional Ventilation in Neonates With Different Delivery Systems of Continuous Positive Airway Pressure
Brief Title: Comparing Different Delivery Systems of Continuous Positive Airway Pressure in Neonates
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jessica E Shui, MD, Neonatologist, Assistant Professor of Pediatrics at MGH, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023P001796
Record Dates: First submitted 2023-08-29; First posted 2023-09-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Prematurity; Respiratory Distress Syndrome
Keywords: continuous positive airway pressure
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Lung physiology measurements with electrical impedance tomography and esophageal manometry will be collected while the participant is supported with RAM cannula ventilator CPAP followed by occlusive interface ventilator CPAP followed by occlusive interface bubble CPAP. A 1:1 block randomization of either A) physiology-based CPAP or B) one size fits all CPAP of either RAM cannula ventilator CPAP or occlusive interface bubble CPAP will be assigned to the participant. Arm B is further randomized 1:1 to either RAM cannula ventilator CPAP or occlusive interface bubble CPAP. The duration of CPAP treatment will be compared between the two arms (precision medicine approach vs standard of care) as well as compare each device and whether the physiology data would have predicted the CPAP device would have resulted in a shorter treatment period.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Given the nature of CPAP, it is not possible to mask which CPAP device the subject is supported by, but the participant, care provider, and outcomes assessor will be masked to whether the subject was randomized to arm A (the device the lung physiology assessment deemed superior for that subject) or arm B (random assignment to the CPAP device, not taking into account the subject's lung physiology).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomization to CPAP with higher change of impedance as measured by EIT. "Arm A-1" (Experimental): After comparing change of impedance as measured by electrical impedance tomography while supported on RAM cannula ventilator CPAP versus occlusive interface bubble CPAP, the participants in this arm are placed on the CPAP that had a greater change of impedance (or less pressure rate product as measured by the esophageal balloon manometry if the change of impedance between the two CPAP modalities are clinically similar).
  In this Arm A-1, these subjects had higher change in impedance while supported on RAM cannula ventilator CPAP
  Interventions: Device: RAM cannula ventilator CPAP
- Randomization to CPAP with higher change of impedance as measured by EIT. "Arm A-2" (Experimental): After comparing change of impedance as measured by electrical impedance tomography while supported on RAM cannula ventilator CPAP versus occlusive interface bubble CPAP, the participants in this arm are placed on the CPAP that had a greater change of impedance (or less pressure rate product as measured by the esophageal balloon manometry if the change of impedance between the two CPAP modalities are clinically similar).
  In this Arm A-2, these subjects had higher change in impedance while supported on occlusive mask bubble CPAP
  Interventions: Device: Occlusive interface bubble CPAP
- Randomization to standard of care - a 'one size fits all' approach. "Arm B-1" (Active Comparator): Currently, the approach to which CPAP modality is chosen for these newborns is defaulted to the preferred CPAP of the Neonatal Intensive Care Unit (NICU) where the newborn is hospitalized.
  In this Arm B-1, these subjects are randomized 1:1 to RAM cannula ventilator CPAP
  Interventions: Device: RAM cannula ventilator CPAP
- Randomization to standard of care - a 'one size fits all' approach. "Arm B-2" (Active Comparator): Currently, the approach to which CPAP modality is chosen for these newborns is defaulted to the preferred CPAP of the NICU where the newborn is hospitalized.
  In this Arm B-2, these subjects are randomized 1:1 to occlusive mask bubble CPAP
  Interventions: Device: Occlusive interface bubble CPAP

INTERVENTIONS:
Device: RAM cannula ventilator CPAP — RAM cannula ventilator CPAP
  Arms: Randomization to CPAP with higher change of impedance as measured by EIT. "Arm A-1"; Randomization to standard of care - a 'one size fits all' approach. "Arm B-1"
Device: Occlusive interface bubble CPAP — Occlusive interface bubble CPAP
  Arms: Randomization to CPAP with higher change of impedance as measured by EIT. "Arm A-2"; Randomization to standard of care - a 'one size fits all' approach. "Arm B-2"

SUMMARY:
The goal of this clinical trial is to compare late preterm newborn lung physiology when supported with different continuous positive airway pressure (CPAP) devices.

The main questions it aims to answer are:

* Which CPAP modality provides better breathing support in newborns with respiratory distress syndrome who are greater than 32 weeks gestational age?
* Does the lung physiology data predict the CPAP modality that will result in a shorter CPAP treatment duration?

Participants will wear a belt of electrodes on their chest (electrical impedance tomography) and have an esophageal balloon manometry measure lung physiology data for 2.5 hours while switching CPAP devices. Participants will then be randomly assigned to a CPAP device to support their breathing until they recover from respiratory distress syndrome.

DETAILED DESCRIPTION:
Across centers, there is a variation in standard of care for the preferred device and interface to deliver continuous positive airway pressure (CPAP) to support neonatal functional residual capacity. CPAP, a type of noninvasive respiratory support, is commonly delivered to neonates by mechanical ventilators or underwater bubble devices (bubble CPAP). Variation also exists with the tubing used to deliver CPAP. One commonly used nasal interface is the RAM cannula (Neotech, Valencia, CA), made of a soft material with thin tubing walls and is designed to provide 60-80% occlusion of the nares. This contrasts with the occlusive interface intended to provide complete seal.

To provide evidence for standardization of CPAP delivery, clinical trials are needed to assess which modality of CPAP delivery is optimal for neonates with respiratory distress syndrome who are > 32 weeks and <37 weeks gestational age, an understudied population. The investigators propose to use electrical impedance tomography (EIT) paired with esophageal balloon manometry to assess neonatal lung physiology when supported with different modalities of CPAP. Furthermore, participants will be randomly assigned to A) physiology based CPAP vs B) one size fits all approach. The subjects will remain on the assigned modality of CPAP for the remainder of their respiratory distress syndrome treatment, and researchers will track which modality of CPAP results in a shorter CPAP treatment period and if this is expected based on the lung physiology data collected.

ELIGIBILITY:
Inclusion Criteria:

* medically stable neonates born >32 0/7 weeks and < 37 0/7 weeks gestational age, with birth weights > 1500 grams, are chronologically 12-36 hours old, and are receiving RAM cannula ventilator CPAP with positive end expiratory pressure (PEEP) between 5-6 cm water (H2O) and Fraction of inspired oxygen (FiO2) < 0.3 for the suspected diagnosis of respiratory distress syndrome

Exclusion Criteria:

* neonates with congenital anomalies that potentially will affect respiratory physiology, for example hypoplastic lungs or gastroschisis.
* neonates with contraindications for wearing an occlusive interface, for example epidermolysis bullosa which may have risk of worsening skin integrity at the pressure points of the occlusive interface, or a known small air leak that may potentially develop into a large pneumothorax.
* neonates with contraindications for placement of esophageal balloon manometry, for example hypoglycemia managed with extended feeding times greater than 30 minutes.
* neonates with contraindications for electrical impedance tomography, for example inability to ensure contact of the electrodes on the belt with the skin on the circumference of the chest due to presence of a chest tube dressing.

Ages: 12 Hours to 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
change in electrical impedance | 2.5 hours during the lung physiology assessment
  change in average electrical impedance with each CPAP delivery modality
duration of CPAP treatment | through study completion, an average of 2 weeks after the lung physiology assessment
  compare groups Arm A-1, A-2 vs Arm B-1, B2; Compare groups Arm A-1, B-1 vs Arm A-2, B-2

SECONDARY OUTCOMES:
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) change in end expiratory lung impedance | 2.5 hours during the lung physiology assessment
  change in end expiratory lung impedance (arbitrary units)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) vascular pulsatility | 2.5 hours during the lung physiology assessment
  vascular pulsatility (arbitrary units)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) tidal volume | 2.5 hours during the lung physiology assessment
  tidal volume (in milliliters) per weight (in kilograms)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) change in minute ventilation | 2.5 hours during the lung physiology assessment
  change in minute ventilation (mL/minute)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) change in dynamic compliance | 2.5 hours during the lung physiology assessment
  change in dynamic compliance (mL/cmH2O)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) Respiratory rate | 2.5 hours during the lung physiology assessment
  Respiratory rate (breaths per minute)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) Oxygen saturation | 2.5 hours during the lung physiology assessment
  Oxygen saturation (percentage)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) Abdominal circumference | 2.5 hours during the lung physiology assessment
  Abdominal circumference (cm)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) esophageal pressure change | 2.5 hours during the lung physiology assessment
  esophageal pressure change (mm Hg)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) end expiratory pressure | 2.5 hours during the lung physiology assessment
  end expiratory pressure via esophageal balloon manometry (mm Hg)
lung physiology measurements (exploratory measures during this pilot study, in preparation for a powered larger trial) pressure rate product | 2.5 hours during the lung physiology assessment
  pressure rate product (cm H2O / min)
clinical outcomes of different CPAP modalities (exploratory measures during this pilot study, in preparation for a powered larger trial) Frequency of deviation | through study completion, an average of 2 weeks after the lung physiology assessment
  frequency of deviation from assigned CPAP treatment (percentage)
clinical outcomes of different CPAP modalities (exploratory measures during this pilot study, in preparation for a powered larger trial) frequency of exogenous surfactant administration | through study completion, an average of 2 weeks after the lung physiology assessment
  frequency of exogenous surfactant administration (percentage)
clinical outcomes of different CPAP modalities (exploratory measures during this pilot study, in preparation for a powered larger trial) | through study completion, an average of 2 weeks after the lung physiology assessment
  respiratory support settings if deviated from assigned CPAP treatment (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica E Shui, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prakash R, De Paoli AG, Davis PG, Oddie SJ, McGuire W. Bubble devices versus other pressure sources for nasal continuous positive airway pressure in preterm infants. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD015130. doi: 10.1002/14651858.CD015130. PMID 37009665
- [Background] Prakash R, De Paoli AG, Oddie SJ, Davis PG, McGuire W. Masks versus prongs as interfaces for nasal continuous positive airway pressure in preterm infants. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD015129. doi: 10.1002/14651858.CD015129. PMID 36374241
- [Background] Green EA, Dawson JA, Davis PG, De Paoli AG, Roberts CT. Assessment of resistance of nasal continuous positive airway pressure interfaces. Arch Dis Child Fetal Neonatal Ed. 2019 Sep;104(5):F535-F539. doi: 10.1136/archdischild-2018-315838. Epub 2018 Dec 19. PMID 30567774
- [Background] Courtney SE, Pyon KH, Saslow JG, Arnold GK, Pandit PB, Habib RH. Lung recruitment and breathing pattern during variable versus continuous flow nasal continuous positive airway pressure in premature infants: an evaluation of three devices. Pediatrics. 2001 Feb;107(2):304-8. doi: 10.1542/peds.107.2.304. PMID 11158463
- [Background] Nascimento MS, do Prado C, Costa ELV, Alcala GC, Correa LC, Rossi FS, Amato MBP, Rebello CM. Effect of flow rate on the end-expiratory lung volume in infants with bronchiolitis using high-flow nasal cannula evaluated through electrical impedance tomography. Pediatr Pulmonol. 2022 Nov;57(11):2681-2687. doi: 10.1002/ppul.26082. Epub 2022 Aug 17. PMID 35931651
- [Background] Seddon PC, Davis GM. Validity of esophageal pressure measurements with positive end-expiratory pressure in preterm infants. Pediatr Pulmonol. 2003 Sep;36(3):216-22. doi: 10.1002/ppul.10284. PMID 12910583
- [Background] Bhatia R, Davis PG, Tingay DG. Regional Volume Characteristics of the Preterm Infant Receiving First Intention Continuous Positive Airway Pressure. J Pediatr. 2017 Aug;187:80-88.e2. doi: 10.1016/j.jpeds.2017.04.046. Epub 2017 May 22. PMID 28545875